CLINICAL TRIAL: NCT04314674
Title: Comparison of Continuous Infusion of 3% Hypertonic Saline, Bolus of 3% Hypertonic Saline and Mannitol on Brain Relaxation During Supratentorial Tumor Resection: A Prospective, Randomized, Clinical Study
Brief Title: Comparison of Hypertonic Saline and Mannitol on Brain Relaxation During Supratentorial Tumors Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Eren Fatma Akcil, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neuroanesthesia Cerrahpasa
Record Dates: First submitted 2020-03-15; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Brain Tumor - Metastatic; Brain Tumor, Adult: Glioblastoma
Keywords: hypertonic saline, mannitol, supratentorial brain tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Mannitol

STUDY DESIGN:
Intervention Model Description: Group 1: %3 HS bolus 3 mL.kg-1 Group 2: %3 HS infusion 20 ml/h Group 3: %20 mannitol 0,6 gr.kg-1
Who Masked: Participant, Investigator
Masking Description: All the patients, the anesthesiologist who will evaluate the postoperative cranial CT will be blind to study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- %3 HS bolus 3 mL.kg-1 (Active Comparator): After the head fixation 3 mL.kg-1 %3 hypertonic saline will be administered over the 20 min intravenously.
  Interventions: Drug: %3 HS bolus
- %3 HS infusion 20 ml/h (Active Comparator): After the head fixation 3% hypertonic saline at 20 ml/h infusion rate will be administered during the operation
  Interventions: Drug: %3 HS infusion 20 ml/h
- %20 mannitol 0,6 gr.kg-1 (Active Comparator): After the head fixation %20 mannitol 0,6 gr.kg-1 will be administered over the 20 min intravenously.
  Interventions: Drug: 20% mannitol

INTERVENTIONS:
Drug: %3 HS bolus — After head fixation %3 HS bolus 3 ml/kg will be administered
  Other Names: Group 1
  Arms: %3 HS bolus 3 mL.kg-1
Drug: %3 HS infusion 20 ml/h — After head fixation %3 HS 20 ml/h infusion will be administered
  Other Names: Group 2
  Arms: %3 HS infusion 20 ml/h
Drug: 20% mannitol — After head fixation %20 mannitol 0.6 ml/kg will be administered
  Other Names: Group 3
  Arms: %20 mannitol 0,6 gr.kg-1

SUMMARY:
Hyperosmotic agents are used to decrease intracranial pressure. The aim of the study is to compare the effects of continuous 3% hypertonic saline (HS), bolus HS and 20% mannitol on intraoperative brain relaxation in patients with raised intracranial pressure during surgery for supratentorial tumors.

DETAILED DESCRIPTION:
After obtaining approval from the ethics committee and informed consent, a total of 90 patients aged 18-70 years, conscious (GCS>13) and American Society of Anesthesiologists (ASA) class I-III, who had intracranial shift >0.5 cm or glioblastoma multiforme or metastatic tumor and who were scheduled for supratentorial mass resection under elective conditions, will be included in the present prospective, randomized, double-blind and placebo-controlled study. Patients with heart failure, kidney insufficiency, diabetes insipidus, electrolyte imbalance and who are unconscious will be excluded from the study.

The patients will randomized into 3 groups:

Group 1: %3 HS bolus 3 mL.kg-1 Group 2: %3 HS infusion 20 ml/h Group 3: %20 mannitol 0,6 gr.kg-1 After head fixation, all patients will be administered with HS or mannitol (over 20 minutes). Arterial blood gas (ABG) analysis (Cobas b 221 blood gas analyzer, Roche®, Basel, Switzerland) will be made at 30 minute,2,4,6,8. hours. Blood sodium, potassium, chlorine, base excess, lactate levels and blood osmolarity will be recorded in each time intervals. The brain relaxation scale will be recorded at the time of dura opening.

ELIGIBILITY:
Inclusion Criteria:

* Elective supratentorial tumor resection
* Glioblastoma multiforme
* Metastatic tumor
* Intracranial shift >0.5 cm
* GCS>13

Exclusion Criteria:

* Renal failure
* Heart failure
* Electrolyte imbalance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Brain relaxation score | 1. min before dura closure
  Brain relaxation score 1: Brain is under the dura, 2: Brain is in the dura level, 3:Brain is above the dura, 4: There is no pulsation in the brain

SECONDARY OUTCOMES:
Sodium level | Baseline and after the drug administration 30. min, 2,4,6,8. hours
  Blood sodium levels obtained from arterial blood gases analysis
Potassium level | Baseline and after the drug administration 30. min, 2,4,6,8. hours
  Blood potassium levels obtained from arterial blood gases analysis

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Tunali, Study Director — Professor of the department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quentin C, Charbonneau S, Moumdjian R, Lallo A, Bouthilier A, Fournier-Gosselin MP, Bojanowski M, Ruel M, Sylvestre MP, Girard F. A comparison of two doses of mannitol on brain relaxation during supratentorial brain tumor craniotomy: a randomized trial. Anesth Analg. 2013 Apr;116(4):862-8. doi: 10.1213/ANE.0b013e318282dc70. Epub 2013 Jan 25. PMID 23354336
- [Background] Dostal P, Dostalova V, Schreiberova J, Tyll T, Habalova J, Cerny V, Rehak S, Cesak T. A comparison of equivolume, equiosmolar solutions of hypertonic saline and mannitol for brain relaxation in patients undergoing elective intracranial tumor surgery: a randomized clinical trial. J Neurosurg Anesthesiol. 2015 Jan;27(1):51-6. doi: 10.1097/ANA.0000000000000091. PMID 25036870
- [Background] Hernandez-Palazon J, Fuentes-Garcia D, Domenech-Asensi P, Piqueras-Perez C, Falcon-Arana L, Burguillos-Lopez S. A comparison of equivolume, equiosmolar solutions of hypertonic saline and mannitol for brain relaxation during elective supratentorial craniotomy. Br J Neurosurg. 2016;30(1):70-5. doi: 10.3109/02688697.2015.1109061. Epub 2015 Nov 16. PMID 26571037